CLINICAL TRIAL: NCT07225751
Title: A Prospective, Randomized, Single-blind, Controlled, Multi-center Study to Assess the Safety and Performance of MagnetOsTM Compared to Autogenous Bone Graft in Patients Undergoing Hindfoot or Ankle Fusions
Acronym: ASTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kuros Biosurgery AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FA-2025-001
Record Dates: First submitted 2025-11-03; First posted 2025-11-10 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2025-12

CONDITIONS: Ankle Arthrodesis or Arthroplasty; Hindfoot Fusion; Ankle Deformity; Ankle Disease; Hindfoot Arthrodesis; Hindfoot Pathologies
Keywords: ankle arthrodesis; hindfoot fusion
MeSH Terms: interventions — Transplantation, Autologous

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MagnetOs (Experimental): Interventions
  * Procedure: Instrumented hindfoot or ankle fusion
  * Device: MagnetOs Putty or MagnetOs Easypack Putty
  Interventions: Device: MagnetOs
- Autograft (Active Comparator): Interventions
  * Procedure: Instrumented hindfoot or ankle fusion
  * Device: Autograft
  Interventions: Other: Autograft

INTERVENTIONS:
Device: MagnetOs — MagnetOs will be used at a volume of approximately 1-5 cc's for the TN, CC and ST joints, and up to 10 cc's for the tibiotalar joint.
  Arms: MagnetOs
Other: Autograft — In this study, the comparator is autograft and will be used at a volume of approximately 1-5 cc's for the TN, CC and ST joints, and up to 10 cc's for the tibiotalar joint.
  Arms: Autograft

SUMMARY:
This is a phase IV post-marketing study for MagnetOs Putty and MagnetOs Easypack Putty. MagnetOs is a synthetic bone graft extender product that is routinely used by surgeon as treatment for hindfoot and ankle disorders.

In this study, MagnetOs Putty and MagnetOs Easypack Putty will be use according to the latest Instructions For Use, standalone in the foot and ankle.

DETAILED DESCRIPTION:
In this study, following a screening period of a maximum of 45 days, approximately 126 patients will receive either MagnetOs Putty/Easypack Putty or autograft in conjunction with rigid hardware (arthrodesis) to treat hindfoot and ankle disorders. They will be randomized (1:1) into one of two treatment groups: standard rigid fixation with MagnetOs Putty/Easypack Putty or local autograft from the calcaneus, distal tibia, or proximal tibia.

They will be followed up at discharge at weeks 2, 6, 12, 24 and 52 post-surgery. The primary endpoint will be analyzed at 24 weeks post-op using CT-scan, and patients will continue follow-up for safety and efficacy for one year post operatively.

In this study, MagnetOs will be applied according to the IFU (Putty) approved in the US, Europe, Middle- East and Australia and Easypack Putty (approved in the US).

The surgical procedures studied in this clinical trial will include rigid hardware fixation and supplemental bone graft/substitute in the following procedures: ankle fusion (tibiotalar), subtalar fusion (talocalcaneal), calcaneocuboid fusion, talonavicular fusion, OR double fusion (any combination of any two of the following: subtalar, talonavicular and calcaneocuboid joints. These procedures will be left to the investigator's discretion.

Radiographs images will be taken at screening, weeks 6, 12, 24 and 52; CT-scans will be taken at weeks 24 and 52 post-op If the patient has a secondary surgical intervention (procedure that adjusts or in any way modifies or removes part of the original implant configuration) at any time after the 6 month visit, the next CT scan will not be necessary. Starting at week 12, all XR images will be weight bearing.

ELIGIBILITY:
Inclusion:

1. Patient is able to read/be read, understand, and provide written informed consent and has signed the IRB approved informed consent.
2. Male or female patient ≥ 18 (considered skeletally mature) up to and including 75 years old
3. Patients requiring one of the following hindfoot fusion procedures, using surgical technique, necessitating rigid hardware fixation and supplemental bone graft/ substitute: ankle fusion (tibiotalar) subtalar fusion (talocalcaneal), calcaneocuboid fusion, talonavicular fusion, OR double fusion (any combination of any two of the following: subtalar, talonavicular and calcaneocuboid joints).
4. Hardware parameters - rigid fixation using screws, plates, staples, nails or a combination.

Exclusion:

1. Expected to need secondary intervention within one year following surgery.
2. Had prior fusion or attempted fusion of the joints to be fused.
3. Patient is not ambulatory.
4. Surgical technique where bone graft is not expected to be used.
5. Conditions at the surgeon's discretion in which general bone grafting is not advisable.
6. Radiographic evidence of fractures or pathologies around the fusion that could negatively impact the fusion process (e.g., growth plate fracture around the fusion or bone cysts).
7. Significant vascular impairment proximal to the graft site.
8. Acute and/or chronic infections in the operated area (soft tissue infections; bacterial bone diseases; osteomyelitis)
9. Pre-existing sensory impairment (e.g. diabetes, Charcot). Diabetics patients with HbA1c greater than 7.0 OR that were not sensitive to the 5.07 monofilament will be excluded.
10. Metabolic disorders know to adversely affect the skeleton (e.g., renal osteodystrophy or hypercalcemia).
11. If intraoperative soft tissue coverage is not planned or possible.
12. Receiving treatment with medication interfering with calcium metabolism (chronic use of glucocorticoid and use high dose NSAIDs 800 mg TID for > the first 6 weeks post-op).
13. Has benign or malignant tumor at the surgical site.
14. Has history or presence of active malignancy (non-invasive skin cancer is allowed).
15. Has known substance abuse, psychiatric disorder, or a condition which, in the opinion of the investigator, may influence the healing or ability to comply with protocol requirements (e.g. prisoners, physically or mentally compromised, etc.).
16. Is involved in active litigation relating to his/her foot and ankle condition.
17. Participation in an investigational study within 30 days prior to surgery for study devices.
18. Patient with body mass index (BMI) > 50.
19. Patient cannot comply with all post-operative evaluation and visits .
20. Any pre-existing condition that the surgeon determines could interfere with the patient's ability to perform objective functional measurements.
21. Women who are or intend to become pregnant within the next 12 months.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic fusion by CT scan | Week 24 post-op
  The primary endpoint is the incidence of fusion at each side by CT analysis as assessed by the independent radiological expert at 24 weeks post-op

SECONDARY OUTCOMES:
Radiographic fusion by CT scan | Week 52
  Joint fusion at Week 52 post-surgery assessed by CT-scans determined by an independent radiological expert panel (IREP) in patients undergoing hindfoot or ankle fusions
Radiographic Fusion by plain radiographs | week 12, week 24, week 52 post-surgery
  Joint fusion at Week 12, Week 24 and Week 52 post-surgery assessed by plain radiographs determined by an independent radiological expert panel (IREP) in patients undergoing hindfoot or ankle fusions
Functional | Screening to Week 2, Week 6, Week 12, Week 24 and Week 52 post-surgery.
  Change in Foot Function Index (FFI) from Screening to Week 2, Week 6, Week 12, Week 24 and Week 52 post-surgery. The score ranging from 0% to 100% indicates the severity of a person's foot issues. A score of 100% indicates worst possible pain, while 0% indicates no pain.
Functional | Screening, Week 2, Week 6, Week 12, Week 24 and Week 52 post-surgery.
  Change in Visual Analog Score (VAS) from Screening to Week 2, Week 6, Week 12, Week 24 and Week 52 post-surgery. 0 no pain and 10 worst pain possible
Functional | Screening, Week 2, Week 6, Week 12, Week 24 and Week 52 post-surgery.
  Change in SF-12 from Screening to Week 2, Week 6, Week 12, Week 24 and Week 52 post-surgery. Where 50 is the average health status for general U.S population. A score above 50 indicates better than average, while a score below 50 suggests below average health.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Steadman Philippon Research Institute, Vail, Colorado
  - Erlanger Orthopaedics, Chattanooga, Tennessee